CLINICAL TRIAL: NCT05027217
Title: Sedation, ANalgesia and Delirium MANagement: a Study of Medical, Surgical, Trauma, and Neuro-intensive Care Patients and a COVID-19 Sub-study.
Brief Title: Sedation, ANalgesia and Delirium MANagement in Intensive Care Unit
Acronym: SAnDMAN
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: PID15072; Trials Group Award 2018 (Other Grant/Funding Number: European Society of Intensive Care Medicine (ESICM))
Record Dates: First submitted 2021-08-13; First posted 2021-08-30 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Critical Illness; Sedation Complication; Intensive Care Unit Delirium; Analgesia; Covid19
Keywords: Intensive Care Unit; Delirium; Sedation; Analgesia; COVID-19
MeSH Terms: conditions — Critical Illness; Agnosia; COVID-19; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard ICU Arm (Main study): We will retrospectively collect data from adults (≥18 years) admitted to a participating ICU prior to the COVID-19 surge in the country, who are invasively mechanically ventilated for more than 12 hours. We will include medical, surgical, trauma and neurological/neurosurgical patients who are COVID-19 negative.
  Interventions: Other: No intervention
- COVID19 ICU arm (COVID-19 sub-study): We will retrospectively collect data from adults (≥18 years) admitted to a participating ICU who are invasively mechanically ventilated for more than 12 hours. We will include data from patients admitted with a confirmed diagnosis of acute respiratory failure due to COVID-19 infection.
  Interventions: Other: No intervention
- Non-COVID19 ICU arm (COVID-19 sub-study): We will retrospectively collect data from adults (≥18 years) admitted to a participating ICU who are invasively mechanically ventilated for more than 12 hours. We will include data from medical, surgical, trauma and neurological/neurosurgical patients who are not admitted for COVID-19.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. Arms are subdivided based on patients' diagnostic status on admission to ICU.

SUMMARY:
Patients with acute severe health problems often need to be admitted to specialised hospital wards called Intensive Care Units (ICUs) where they can receive emergency treatment such as mechanical ventilation to support their breathing function via a machine, and sedative medications to reduce pain and anxiety associated with the severity of their condition.

Although these interventions and treatments are often necessary to support patients' vital functions, they also carry the risk of important side effects.

Sedative drugs use in particular, has a significant impact on short- and long-term outcomes.

Despite international guidelines to help clinicians in the use of these drugs, there appears to be large variability in their use around the world such as use of different types of drugs, variable doses or rate of continuous infusions, etc.

However, even with this known variable practice across the world, there are no large-scale international studies looking at the use of sedative drugs, pain-relief medications and drugs to control agitation and restlessness in ICUs.

Therefore, the investigators propose a multinational study to better understand how different ICUs use these drugs and if they follow the guidance published by expert clinicians. The investigators will collect data in more than 100 ICUs across the world and include more than 2000 adult patients admitted to ICU and needing mechanical breathing.

There are no active interventions on patients that are part of this research study and data collection from patients medical records is retrospective. All patients included will receive the standard of care as per their local intensive care unit.

Also, in a 2-arm sub-study, the investigators will collect retrospective data from medical records of patients admitted to ICU before and during the COVID-19 pandemic to explore how sedation, analgesia and delirium practice has changed during this exceptional timeframe.

DETAILED DESCRIPTION:
Study design: Multicentre Retrospective Observational Cohort Study with two-arm COVID-19 sub-study (same design)

ELIGIBILITY:
Inclusion Criteria

Main study

Data will be collected from patients who fulfil all the following inclusion criteria:

1. Standard ICU arm:

* All male or female aged ≥18 years admitted to a participating Intensive Care Units who are invasively mechanically ventilated for more than 12 hours will be included.
* Patients admitted with medical, surgical, trauma, burns, neurological and neurosurgical clinical problems.
* Admitted to ICU prior to the COVID-19 surge in the specific country.

COVID-19 sub-study

Data will be collected from patients who fulfil all the following inclusion criteria:

1. COVID-19 ICU arm:

   * All male or female aged ≥18 years admitted to a participating Intensive Care Units who are invasively mechanically ventilated for more than 12 hours will be included.
   * Patients admitted with pneumonia and/or acute respiratory failure and a diagnosis of COVID-19.

     * The accepted criteria for the diagnosis to COVID-19 includes one of the following: 1) RT-qPCR is positive for SARS-CoV19 nucleic acid; 2) the viral gene identified by gene sequencing; or 3) presence of COVID-19-specified IgM and IgG antibodies.
2. Non-COVID-19 ICU arm:

   * All male or female aged ≥18 years admitted to a participating Intensive Care Units who are invasively mechanically ventilated for more than 12 hours will be included.
   * Patients admitted with medical, surgical, trauma, burns, neurological and neurosurgical clinical problems.
   * No confirmed or suspected COVID-19 disease.

Exclusion Criteria

Main study

Data will not be collected from patients who fulfil the following exclusion criteria:

1. Standard ICU arm:

• Patients admitted to non-acute care units

COVID-19 sub-study

Data will not be collected from patients who fulfil the following exclusion criteria:

1. COVID-19 ICU arm:

   * Patients with confirmed diagnosis of COVID-19 but admitted to ICU for indications different than pneumonia and/or acute respiratory failure (incidental positive COVID-19)
   * Patients admitted to non-acute care units
2. Non-COVID-19 ICU arm:

   * Patients admitted to non-acute care units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to ICU and mechanically ventilated for at least 12 hours.
Sampling Method: Probability Sample
Enrollment: 3421 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Sedation practice | First 7 days of mechanical ventilation
  Number of patient/days for each sedative and analgesic (propofol, benzodiazepines, opioids, etc.).
  Note: a full list of sedatives and analgesics is available in the eCRF.
Use of Pain, Analgesia and Delirium assessments | First 7 days of mechanical ventilation
  Number of patient/days when a Pain, Analgesia and Delirium assessment (any) has been used.
  Note: a list of PAD assessments is available in the eCRF.

SECONDARY OUTCOMES:
Adherence to PADIS guidelines | First 7 days of mechanical ventilation
  Percentage of patient/days with sedation, analgesia and delirium practice compliant to PADIS guidelines.
  Note: The full PADIS recommendations are available at https://pubmed.ncbi.nlm.nih.gov/30113371/
Sedation practice in different cohorts | First 7 days of mechanical ventilation
  Number of patient/days for each sedative/analgesic drug (propofol, benzodiazepines, opioids, etc.) in different subgroups (sepsis and acute respiratory distress syndrome (ARDS), COVID-19, surgical patients, trauma and burns patients, neurocritical care patients, cardiogenic shock patients, patients receiving palliative care).
  Note: a full list of sedatives and analgesics is available in the eCRF.
Delirium | First 7 days of mechanical ventilation
  Number of patient/days when delirium was assessed (any assessment). Number of patient/days receiving treatment for delirium symptoms.
  Note: a full list of delirium assessments and treatment options are available in the eCRF.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Mehta, Prof, Principal Investigator — Sinai Health, Toronto (Canada)
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
SANDMAN investigators will be given priority to lead secondary analyses and are encouraged to do so. Participation and authorship opportunities will be based on contribution to the primary study. The study steering committee will consider the scientific validity and the possible effect on the anonymity of participating centres prior to granting any such requests. Where necessary, a prior written agreement may be requested to set out the terms of such collaborations. Investigators should submit a secondary study proposal for review by the Executive committee. 'Cleaned' data from the international or national datasets will only be released after a secondary study proposal has been approved. An analysis involving any data derived from the SANDMAN study will be considered a secondary analysis and subject to these rules.
Supporting Information: Study Protocol, SAP
Time Frame: After the main study report is published.
Access Criteria: Upon request to the study Executive Committee
URL: https://www.esicm.org/sandman/

REFERENCES:
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Chanques G, Constantin JM, Devlin JW, Ely EW, Fraser GL, Gelinas C, Girard TD, Guerin C, Jabaudon M, Jaber S, Mehta S, Langer T, Murray MJ, Pandharipande P, Patel B, Payen JF, Puntillo K, Rochwerg B, Shehabi Y, Strom T, Olsen HT, Kress JP. Analgesia and sedation in patients with ARDS. Intensive Care Med. 2020 Dec;46(12):2342-2356. doi: 10.1007/s00134-020-06307-9. Epub 2020 Nov 10. PMID 33170331
- [Background] Tanios M, Nguyen HM, Park H, Mehta S, Epstein SK, Youssef F, Beltran A, Flores G, Sidhom R, Sehgal A, Leo J, Devlin JW. Analgesia-first sedation in critically ill adults: A U.S. pilot, randomized controlled trial. J Crit Care. 2019 Oct;53:107-113. doi: 10.1016/j.jcrc.2019.06.008. Epub 2019 Jun 12. PMID 31228760
- See also: ESICM Trials Group - Study documents — https://www.esicm.org/sandman/